CLINICAL TRIAL: NCT06572540
Title: Transthoracic Versus Transbronchial Cryoablation for Early-stage Peripheral Lung Cancer: A Prospective, Randomized Controlled Trial
Brief Title: Transthoracic vs Transbronchial Cryoablation for Early-stage Peripheral Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiayuan Sun (Other)
Responsible Party: Sponsor-Investigator, Jiayuan Sun, Director, Department of Respiratory Endoscopy, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AT-RXLD-202401
Record Dates: First submitted 2024-08-20; First posted 2024-08-27 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer
Keywords: Cryoablation; Lung cancer; Transbronchial ablation; Transthoracic ablation
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transthoracic cryoablation (Active Comparator): Subjects will undergo CT-guided cryoablation. According to the location of the lesion on the chest CT scan, the puncture point, direction of needle entry, and distance of needle entry will be determined. The primary cryoablation needle (via the chest wall) will be punctured into the lesion according to the pre-planed path, and the CT will confirm the correct position. One or more needles will rationally distributed in the lesion for ablation according to the morphology of the lesion.
  Interventions: Device: Transthoracic cryoablation
- Transbronchial cryoablation (Experimental): Subjects will undergo bronchoscopically guided cryoablation. Appropriate guided bronchoscopic technique will be uesd. Cryoablation needle (flexible) will insert through the working channel of the bronchoscope to the target lesion, CBCT will be used to confirm the correct position and observe the ablation zone.
  Interventions: Device: Transbronchial cryoablation

INTERVENTIONS:
Device: Transthoracic cryoablation — Transthoracic cryoablation will be performed under the guidance of CT.
  Arms: Transthoracic cryoablation
Device: Transbronchial cryoablation — Transbronchial cryoablation will be performed under the guidance of navigation bronchoscopy and CBCT.
  Arms: Transbronchial cryoablation

SUMMARY:
The study aims to compare the efficacy and safety of transthoracic cryoablation to transbronchial cryoablation in the treatment of early-stage peripheral lung cancer.

DETAILED DESCRIPTION:
Ablation therapy has been widely used in the treatment of peripheral lung cancer. Among various ablation techniques, cryoablation has been demonstrated to be therapeutic efficacy with several advantages, including high safety, clear ablation borders, and minimal local pain. With the development of navigational bronchoscopy, pilot study on transbronchial cryoablation for peripheral lung cancer has proved its efficacy and safety, but there is a lack of prospective randomized controlled trials to verify its near-term as well as long-term efficacy and safety. This study was designed as a prospective, randomized controlled, multicenter clinical trial. A total of 110 participants will be randomly assigned to either the transbronchial group or the transthoracic group in a 1:1 ratio. The primary endpoint is the complete ablation rate at 12 months post-ablation. Secondary endpoints include technical success rate, complete ablation rate at 6 months post-ablation, local control rate at 1, 2 and 3 years post-ablation, progression-free survival, overall survival, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 18 years.
2. Primary peripheral lung cancer diagnosed by pathology and pre-procedure staging examination suggesting clinical stage T1N0M0, stage IA (including postoperative new and multiple primary).
3. The target lesion was evaluated to be feasible for both CT and bronchoscopy-guided ablation.
4. Patients who are not suitable for surgery or refuse surgery, agree to undergo initial ablation therapy and sign informed consent form.

Exclusion Criteria:

1. Patients with platelets <70×109/L, severe bleeding tendency and coagulation dysfunction that cannot be corrected in a short term.
2. Patients with severe pulmonary fibrosis and pulmonary arterial hypertension.
3. Infectious and radioactive inflammation around the lesion, skin infection at the puncture site that is not well controlled, systemic infection, high fever >38.5°C.
4. Patients with severe hepatic, renal, cardiac, pulmonary and cerebral insufficiency, severe anaemia, dehydration and serious disorders of nutritional metabolism that cannot be corrected or improved in a short term.
5. Those with poorly controlled malignant pleural effusions.
6. Anticoagulation therapy and/or anti-platelet drugs (except dabigatran, rivaroxaban and other new oral anticoagulants) have not been discontinued more than 5~7d before ablation.
7. Eastern Cooperative Oncology Group (ECOG) score >2.
8. Combination with other tumors with extensive metastases and an expected survival of <6 months.
9. Patients with episodic psychosis.
10. Pregnant women, or patients with pregnancy plan during the study period.
11. Have participated or are participating in other clinical studies within 30 days.
12. Any other condition that the investigator considers inappropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete ablation rate at 12 months | Twelve months post-ablation
  Twelve months after the overall ablation procedure, the proportion that subjects whose lesion recevied ablation maintain completely ablated account for all evaluable subjects who receive cryoablation.

SECONDARY OUTCOMES:
Technical success rate | Immediately after Each Operation
  It is defined as the number of lesions for which the ablation needle reached the location of the lesion and was successfully ablated as a proportion of the total number of lesions to be ablated, as assessed by immediate post-ablation imaging
Complete ablation rate at 6 months | Six months post-ablation
  Six months after the overall ablation procedure, the proportion that subjects whose lesion recevied ablation maintain completely ablated account for all evaluable subjects who receive cryoablation.
Local control rates at 1, 2 and 3 years postoperatively | 12, 24, 36 monthspost-ablation
  The number of lesions with complete and incomplete ablation at 1, 2, and 3 years after ablation treatment as a proportion of the number of all ablation-treated lesions.
Progression-free survival (PFS) | From the time of treatment to the time of disease progression or death (determined by the one which occurs first), up to 36 months
  PFS was defined from the first day after ablation to progression of target lesions and/or appearance of new lesions or death.
Overall survival（OS） | From the time of treatment to the time of the patient death, up to 36 months
  Overall survival（OS) is evaluated after the treatment of ablation until the patient death.
Adverse event | Twelve months psot-ablation
  All adverse events will be recorded during operation and during the follow-up, and be evaluated according to the CTCAE v5.0. Related and possible related AEs and SAEs will be determined and evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, PhD, Study Director — Shanghai Chest Hospital
Locations (5):
- China (5):
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Shanghai Chest Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital , affiliated with the Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No